CLINICAL TRIAL: NCT00974558
Title: The Use of a Handheld Fan to Improve Breathlessness - a Feasibility Study to Assess Relief From Breathlessness After Five Minutes Use of a Handheld Fan Directed at the Cheeks
Brief Title: The Use of a Handheld Fan to Manage Breathlessness - A Feasibility Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Collaborators: St Catherines Hospice (Unknown); Scarborough acute hospitals Trust (Unknown); University hospitals Morecambe Bay (Unknown); St Johns Hospice (Unknown)
Responsible Party: Principal Investigator, Sarah Galbraith, Consultant in palliative medicine, Cambridge University Hospitals NHS Foundation Trust
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A091619
Record Dates: First submitted 2009-09-09; First posted 2009-09-10 (Estimated); Last update posted 2015-02-02 (Estimated); Status verified 2015-01

CONDITIONS: Dyspnea
Keywords: dyspnea; fan
MeSH Terms: conditions — Dyspnea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- fan directed to cheeks (Experimental): Blow draft of air generated by fan across cheeks
  Interventions: Device: handheld fan directed to cheeks

INTERVENTIONS:
Device: handheld fan directed to cheeks — Handheld fan directed to cheeks for 5 minutes
  Other Names: handheld fan

SUMMARY:
The aim of the study is to investigate if the use of a handheld fan directed to the cheeks alongside conventional medical treatment partially or totally relieves breathlessness and if this effect lasts for at least 30 minutes in patients irrespective of the underlying disease process.

DETAILED DESCRIPTION:
A previous randomised controlled trial (Galbraith et al, accepted for publication) has shown a reduction in breathlessness after 5 minutes use of a fan directed to the cheeks. This study is a feasibility study to determine how long this beneficial effect lasts.

With the patient in a relaxed sitting position and ensuring there is no other fan or open window blowing air onto the subject, the following will be explained to the patient and then measured and recorded

* Numerical Rating Scale (NRS) for dyspnoea
* Visual analogue scale (VAS) for breathlessness with end anchors
* O2 saturation using pulse oximeter
* Pulse rate using pulse oximeter
* Room temperature and humidity recorded

The patients will be asked to avoid talking or significantly change position throughout the study.

Fan to cheeks The investigator will demonstrate to the patient how to use the handheld fan directed to the cheeks. The appropriate area on the face, which corresponds to the area innervated by 2nd and 3rd trigeminal nerve branches, will be demonstrated by the researcher. The patient will then use the fan as demonstrated and this will be timed for 5 minutes with the patient in a relaxed sitting position.

Assessment following treatment with fan After 5 minutes use of the fan directed at cheeks, the following will be recorded immediately

* NRS and VAS for dyspnoea
* Relief score, a 5 point rating of how much relief from breathlessness the participant has obtained (0=nil, 1= a little relief , 2= moderate relief, 3=good relief, 4=no longer breathless/maximal relief)
* O2 saturation
* Pulse rate

Participants who have had no improvement in breathlessness as measured by VAS, NRS or gained no relief assessed by the relief score will end the study at this point.

Participants who have an improvement in breathlessness will continue the study and NRS and VAS will to be recorded every 10 minutes in alternating order until the NRS or/and VAS have returned to baseline values or reached a steady level.

ELIGIBILITY:
Inclusion Criteria:

* Any patient able and willing to cooperate with the study and who defines themselves as breathless at rest by answering 'yes' to the question, 'Do you currently feel short of breath?'
* Any diagnosis causing breathlessness
* Age >3 0years

Exclusion Criteria:

* Patients who have previously used a handheld fan to manage their breathlessness
* Patients with fever >38 0C in last 24 hours
* Patients on continuous oxygen
* Patients requiring short burst oxygen therapy whilst completing the study
* Patients with diseases or treatment affecting the trigeminal nerve supply.
* Patients with other diseases which, in the opinion of the researcher or investigator, may affect the mechanism of action of the fan
* Patients unable to understand or cooperate with study
* Patients who do not wish to participate in the study

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2010-01; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
Primary outcome measure is time in minutes for which breathlessness is improved after 5 minutes use of the fan directed at the face | 2 hours

SECONDARY OUTCOMES:
Relief from breathlessness noted on relief score after using the handheld fan | 2 hours
Correlation between VAS and NRS scales | 2 hours

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Galbraith, BM, Principal Investigator — Cambridge UNiversity Hospitals NHS Foundation Trust Addenbrookes Hospital; Sara Booth, MD, Study Director — Cambridge University Hospitals NHS Foundation Trust Addenbrookes Hospital
Locations (1):
- Addenbrookes Hospital, Cambridge, Cambs, United Kingdom